CLINICAL TRIAL: NCT02847247
Title: Systemic Inflammatory Response to 20,000 EU Clinical Center Reference Endotoxin in Normal Adults
Brief Title: Systemic Inflammatory Response to CCRE
Acronym: Endoscreen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-1458
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Healthy
Keywords: healthy
MeSH Terms: interventions — Endotoxins; Lipopolysaccharides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CCRE (Experimental): 20,000 EU of CCRE (Clinical Center Reference Endotoxin)
  Interventions: Drug: CCRE

INTERVENTIONS:
Drug: CCRE — Endotoxin challenge: Subjects will undergo inhalation of 20,000 EU CCRE. The CCRE will be inhaled by subjects as a nebulized preparation using an ultrasonic nebulizer until the challenge solution is completely spent (generally 10 minutes).
  Other Names: endotoxin, lipopolysaccharide (LPS)

SUMMARY:
Purpose: The purpose of this study is to classify volunteers as endotoxin-responders or non-responders following inhalation of 20,000 EU Clinical Center Reference Endotoxin (CCRE). Endotoxin is a commonly encountered bioaerosol and component of indoor and outdoor air pollution. For reasons that remain unclear, some individuals appear to be more susceptible to the inflammatory effects of inhaled endotoxin than are others, possibly owing to single nucleotide polymorphisms in the Toll-like receptor 4 (TLR4) gene that influence TLR4 signaling and function. These susceptible individuals represent a population of particular interest for further mechanistic studies of the effects of endotoxin and for therapeutic trials. Susceptibility to inhaled endotoxin will be determined by measuring change in peripheral blood neutrophil counts, a biomarker of systemic inflammation, following inhaled CCRE. In our previous work, the investigators have found that inhalation of 20,000 EU CCRE is well tolerated and induces measurable increase in neutrophil content of peripheral blood in susceptible individuals. Our hope is that this CCRE inhalation protocol can be employed to screen large populations for susceptibility to the inflammatory effect of inhaled endotoxin.

DETAILED DESCRIPTION:
This is a single center, screening study involving recruitment of 18 normal volunteers (NV). The protocol is powered to compare absolute neutrophil count (ANC) in the blood 6 hours after inhalational challenge with CCRE compared baseline. In addition, as secondary endpoints, the investigators will evaluate inflammatory cytokine levels in systemic circulation and access for the presence of genes thought to be related to endotoxin response. Visits will be conducted by a study coordinator or other study staff, physical exams will be performed by the PI or other study physician.

Eighteen subjects will be recruited. There will be no gender or ethnic restrictions, and subjects will be healthy volunteers. Prior to enrollment in this study, subjects will have participated in our protocol 98-0799 (screening and database study for the CEMALB). Data such as medical history and allergy skin testing collected during the screening protocol will be included with data in this study. Subjects with positive allergy skin testing will not be excluded. Spirometry will be performed to determine the current level of lung function.

In order to identify those individuals who appear more susceptible to the systemic inflammatory effects of endotoxin exposure, subjects will undergo inhaled endotoxin challenge at the baseline visit followed 6 hours later by blood draw for complete blood count with differential to allow for calculation of absolute neutrophil count (ANC). Subjects will be considered "responders" if their peripheral ANC increases by at least 20% following inhaled endotoxin challenge.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18-50 years of age to be eligible for study participation
2. Subjects must be willing to and able to provide informed consent and participate in all study procedures
3. Normal lung function, defined as (Knudson 1976/1984 predicted set):

   * 1. Forced Vital Capacity (FVC) of > 80% of that predicted for gender, ethnicity, age and height
   * 2. Forced Expiratory Volume in the first second (FEV1) of > 80% of that predicted for gender, ethnicity, age and height
   * 3. FEV1/FVC ratio of > 0.75 of that predicted for gender, ethnicity, age and height
4. Oxygen saturation of > 94% Normal blood pressure (Systolic between 150 - 90, Diastolic between 90-60 mm Hg)
5. Symptom Score (defined in section "f") no greater than 6 (out of a possible 24) for total symptom score with a value no greater than 2 for any one score.

Exclusion Criteria:

1. Any chronic medical condition considered by the PI as a contraindication to the exposure study including significant cardiovascular disease, diabetes requiring medication, chronic renal disease, or chronic thyroid disease.
2. Physician directed emergency treatment for asthma exacerbation within the preceding 3 months.
3. Moderate or Severe asthma
4. Exacerbation of asthma more than 2x/week that would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
5. Nighttime symptoms of cough or wheeze greater than 1x/week at baseline (not during a clearly recognized viral induced asthma exacerbation) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma
6. Daily requirement for albuterol due to asthma symptoms (cough, wheeze, chest tightness) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma. (Not to include prophylactic use of albuterol prior to exercise).
7. History of intubation for asthma
8. Daily use of NSAIDs, or inability to withhold NSAIDs for 4 days prior to dosing.
9. Use of medications that may impact the results of the study to include, but not limited to, systemic corticosteroids, beta blockers.
10. Cigarette smoking > 1 pack per month.
11. BMI>35.
12. Pregnant or breast feeding women will not be included.
13. Subjects who are employed within the past 6 months in an occupation with high risk for endotoxin exposure, such as grain storage sites or swine containment.
14. Subjects will be deferred after any acute, non-chronic medical condition requiring treatment, such as bronchitis, pneumonia or febrile illness for a minimum of 4 weeks after complete resolution of symptoms.

    -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
Change in peripheral blood PMNs | 6 hrs post exposure
  The objective of this study is to identify endotoxin responders, characterized by an increase in post-CCRE peripheral blood polymorphonuclear (PMN)s compared to that day's baseline values of > 20%. Thus, there will be two data points for this cohort, blood PMNs at baseline and PMNs 6 hours following 20,000 endotoxin units (EU) of CCRE.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hernandez, MD, Principal Investigator — UNC
Locations (1):
- Environmental Protection Agency Human Studies facility, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
for internal analysis only